CLINICAL TRIAL: NCT04197869
Title: Does a Preoperative Bowel Regimen Change Time to First Bowel Movement After Robotic Sacral Colpopexy: A Randomized Controlled Trial
Brief Title: Does a Preoperative Bowel Regimen Change Time to First Bowel Movement After Robotic Sacral Colpopexy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0802
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Constipation; Post-Op Complication
MeSH Terms: conditions — Constipation; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: The experimental group will take a pre-operative course of polyethylene glycol daily for seven days prior to procedure date. The control group will not be given any intervention preoperatively. All patients will take polyethylene glycol postoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will take a pre-operative course of polyethylene glycol daily for seven days prior to procedure date.
  Interventions: Drug: Polyethylene Glycol Powder
- Control (No Intervention): The control group will not be given any intervention preoperatively.

INTERVENTIONS:
Drug: Polyethylene Glycol Powder — Polyethylene Glycol 3350 17g should be mixed in 8 ounces of fluid for administration. Polyethylene glycol is a high molecular weight, water soluble polymer which can form hydrogen bonds with water molecules. It is an osmotic laxative solution which stimulates bowel movements by increasing the amount of water absorbed in the GI tract. It decreases feces consistency and increases their volume by promoting peristalsis and evacuation. The side effects of polyethylene glycol are bloating, gas or diarrhea. The half-life of polyethylene glycol is 4-6 hours and after 18 hours the concentration declines to non-quantifiable levels.
  Arms: Experimental

SUMMARY:
The hypothesis is that starting a bowel regimen with Polyethylene Glycol prior to robotic assisted sacrocolpopexy will decrease time to first bowel movement after surgery. The experimental group will take a pre-operative course of polyethylene glycol daily for seven days prior to procedure date. The control group will not be given any intervention preoperatively. All patients will take polyethylene glycol postoperatively.

DETAILED DESCRIPTION:
In order to assess bowel characteristics and assess for pre-existing constipation a standardized questionnaire will be distributed to all patients prior to surgery at their pre-operative visit. The patients in the experimental group will have follow up via phone call, 3-4 days prior to surgery to assess for medication compliance or any side effects/complications. Patients will record if they are taking their Miralax as prescribed daily. They will also record their bowel movements and pain levels during evacuation. Prior to surgery, in the pre-operative area, medication compliance will be assessed once again. Post operatively all patients will take polyethylene glycol for seven days, once a day. They will maintain a bowel diary, which will record bowel movements, stool type and pain with evacuation. The primary objective is to determine if the preoperative use of polyethylene glycol decreases time to first bowel movement after robotic sacral colpopexy. Secondary outcomes include pain with first bowel movement, stool consistency and daily pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a robotic assisted sacrocolpopexy with or without hysterectomy and with or without anti-incontinence procedures

Exclusion Criteria:

* Age under 18 or over 90
* Planned laparotomy
* Planned posterior colporrhaphy
* Regular pre-operative use of stool softeners/laxatives
* Presence of colostomy
* Inability to give informed consent
* Inability to take medication by mouth
* Chronic kidney disease (Cr > 1.2)
* Esophageal strictures
* Persistent nausea and vomiting
* Bowel obstruction
* Inflammatory bowel disease

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Bay Shore, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holubyeva A, Goodwin AI, O'Shaughnessy D, Pillalamarri N, Demertzis K, Rahbani AC, Stefanov DG, Finamore PS. Does a Preoperative Bowel Regimen Change Time to Bowel Movement? A Randomized Clinical Trial. Urogynecology (Phila). 2024 Mar 1;30(3):251-255. doi: 10.1097/SPV.0000000000001462. Epub 2024 Feb 26. PMID 38484239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Control
Started | 34 | 37
Completed | 24 | 25
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.8) | 60.4 (8.7) | 62.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 2
  Hispanic or Latino | 2 | 2 | 4
  White | 21 | 21 | 42
  Unknown/not reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: First Bowel Movement
Description: Time to first post-operative bowel movement will be evaluated.
Time Frame: 7 days post-operatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 24 | 25
days | 1.96 (1) | 2.32 (0.99)

2. Secondary Outcome: Post Operative Pain With First Bowel Movement as Measured by the VAS Scale.
Description: Patients will record their pain levels with first post-operative bowel movement using the Visual Analogue Scale (VAS) pain scale. The scale is numbered 0 through 10, with 0 being no pain and 10 being worst possible pain.
Time Frame: 7 days post-operatively
Population: one experimental patient did not report this data point therefore there were 23, not 24, patients analyzed
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 23 | 25
units on a scale | 1 [0 to 2] | 4 [2 to 5]

3. Secondary Outcome: Post Operative Pain at Day 1 as Measured by the VAS Scale
Description: Patients will record their pain level using the Visual Analogue Scale (VAS) pain scale. The scale is numbered 0 through 10, with 0 being no pain and 10 being worst possible pain.
Time Frame: 1 day post-operatively
Population: Some patients did not report this data point therefore there were fewer patients analyzed than were described in the Participant Flow
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 18 | 21
units on a scale | 4 [3 to 6] | 2 [0 to 4]

4. Secondary Outcome: Median Postoperative Pain
Description: Patients will record their pain level daily for 7 days using the Visual Analogue Scale (VAS) pain scale. The scale is numbered 0 through 10, with 0 being no pain and 10 being worst possible pain. The average value over 7 days for each patient will be calculated. We will then report the median postoperative pain score averaged across 7 days for each group.
Time Frame: Averaged over 7 days post-operatively
Population: One patient did not report this data point therefore there were fewer patients analyzed than were described in the Participant Flow
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 23 | 25
units on a scale | 1.3 [0 to 2.9] | 3.2 [2.3 to 3.6]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 month
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 3/24 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=24) | Control (N=25)
loose stool (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT04197869/Prot_SAP_000.pdf